CLINICAL TRIAL: NCT02188810
Title: A Phase I Randomized, Observer-blind, Controlled, Dose Escalation Trial of the Safety and Tolerability of a Single Intramuscular Dose of a PAL Adjuvant (FB-631) Co-administered With Seasonal TIV (2013-2014) in Healthy Adults.
Brief Title: Safety and Reactogenicity of a PAL Combined With Seasonal Flu Vaccine in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Folia Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PE1202
Record Dates: First submitted 2014-07-01; First posted 2014-07-14 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Flu
Keywords: PAL; fluviral; healthy volunteer; adjuvant; TH1 immune response
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Active Comparator): Single dose of control vaccine (a single dose of 0.5 mL TIV).
  Interventions: Biological: TIV
- Group 2 (Experimental): Single dose of the test article (0.25 mL TIV, which is 7.5 μg of each influenza strain with 0.5x PAL, i.e. 30 μg).
  Interventions: Biological: PAL; Biological: TIV
- Group 3 (Experimental): Single dose of the test article (0.25 mL TIV, which is 7.5 μg of each influenza strain with 1x PAL, i.e. 60 μg).
  Interventions: Biological: PAL; Biological: TIV
- Group 4 (Experimental): Single dose of the test article (0.25 mL of TIV which is 7.5 μg of each influenza strain with 2x PAL (i.e., 120 μg).
  Interventions: Biological: PAL; Biological: TIV
- Group 5 (Experimental): Single dose of the test article (0.25 mL of TIV which is 7.5 μg of each influenza strain with 4x PAL (i.e., 240 μg).
  Interventions: Biological: PAL; Biological: TIV
- Group 6 (Experimental): Single dose of the test article (0.125 mL of TIV with 4x PAL i.e., 240 μg).
  Interventions: Biological: PAL; Biological: TIV

INTERVENTIONS:
Biological: PAL — Single dose administered intramuscularly.
  Other Names: PapMV Adjuvant Long lasting immune response; FB-631
  Arms: Group 2; Group 3; Group 4; Group 5; Group 6
Biological: TIV — Single dose administered intramuscularly .
  Other Names: Trivalent Influenza Vaccines; Fluviral

SUMMARY:
This is a phase 1, research study is looking at the safety and acceptability of a new vaccine adjuvant (immune booster) called PAL when combined with the seasonal flu vaccine (Fluviral) to test the safety and effectiveness of new vaccines and medications on healthy volunteers.

The study will enroll approximately 48 healthy adult participants, and occur over 3 years. In the first six months/180 days of the study participants will have visits to the study site during which safety and immunogenicity outcomes will be measured. From Day 181 to Year 3, participants will be contacted by telephone or email to collect information on any adverse events.

DETAILED DESCRIPTION:
This is a phase 1, dose-ranging, randomized (5:1), observer-blind, controlled study of the safety and immune response to intramuscular injection of PapMV (Papaya Mosaic Virus) rVLP (Recombinant Virus-Like Particles) which is PAL adjuvant, or "PAL" combined with Trivalent Influenza Vaccines (TIV) at one of four dose levels of PAL, combined with one of two dose levels of TIV, or active control (TIV). The study will enroll approximately 48 healthy adult participants, and occur over 3 years. In the first six months/180 days (Epoch 1) of the study participants will have visits to the study site during which safety and immunogenicity outcomes will be measured. In Epoch 2 (Day 181 to Year 3) participants will be contacted by telephone or email to collect unsolicited adverse events.

This is a controlled clinical trial. The control group will receive the standard dose of TIV, 0.5 mL, which consists of 15 μg haemagglutinin (HA) of each influenza strain recommended by the World Health Organization (WHO) for the 2013-2014 influenza season in the northern hemisphere. An active control is used so that the attributable risk of adverse events can be estimated, and so that outcome measures can be assessed in a blinded fashion. Only adults in stable health will be eligible in order to minimize participant risk. Only non-pregnant females of childbearing age are eligible, and they must agree to continue adequate contraception for 180 days after injection. Study holding rules and a safety evaluation by a Safety Review Committee (SRC) will be in place. The study will follow a staggered dose-escalation design, with each of four steps introducing a new dose of the adjuvant (30, 60, 120 and 240 μg respectively).

The first dose level of PAL adjuvant FB-631 is 0.5 X 60 µg (i.e., 30 µg), which is half the dose that was found to be most immunogenic in animal studies. The adjuvant is co-administered with 0.25 mL of TIV, which is half the dose of TIV that is routinely administered to adults (i.e. 7.5 μg of each of the three influenza subtypes contained in the vaccine). The next dose level is 60µg of FB-631 combined with 0.25 mL TIV. The third dose level is 120 μg of FB-631 with 0.25 mL TIV. In the fourth and final step the dose of adjuvant is 240 μg of PAL adjuvant combined with 0.25 mL TIV (8 participants) or 0.125 mL TIV (i.e. 3.75 μg HA of each influenza subtype contained in the vaccine) (8 participants).

Any safety signal observed in the study will lead to a hold until the decision of Safety Review Committee to continue, modify or suspend the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

* Good general health status, as determined by history and physical examination no greater than 30 days prior to administration of the first test article.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of Diary Cards, return for follow-up visits).
* If female of child-bearing potential and heterosexually active, has practiced adequate contraception for 30 days prior to injection and has a negative pregnancy test on the day of injection and has agreed to continue adequate contraception until 180 days after injection. (Please refer to the glossary for the definition of child-bearing potential and adequate contraception).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study product within 28 days preceding the dose of study product, or planned use during the study period.
* Planned administration/ administration of a vaccine/product not foreseen by the study protocol within the period starting 28 days before injection and ending 28 days after.
* Planned administration/ administration of the seasonal influenza vaccine recommended by local public health authorities within the period starting 120 days before injection and ending 121 days after. (Note: enrolment should be completed 120 days before the annual seasonal influenza vaccine campaigns in October and December)
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study product or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination. (Laboratory testing for HIV, Hepatitis C and Hepatitis B will be performed during the screening visit).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drug within 6 months prior to the product dose
* Family history of congenital or hereditary immunodeficiency.
* History of or current autoimmune disease.
* Known or suspected hypersensitivity to Fluviral, to thimerosal, or to any other ingredient in the formulation or component of the container.
* Pregnant or lactating female.
* Any hematological (hemoglobin level, white blood cell [WBC], and platelet count) and biochemical (alanine aminotransferase [ALT], aspartate aminotransferase [AST], blood urea nitrogen [BUN] and creatinine) abnormality as per local laboratory normal values considered clinically significant by the investigator.
* Any acute or chronic, clinically significant disease, as determined by physical examination or laboratory screening tests.
* Any other condition that the investigator judges may interfere with study procedures (e.g. drawing blood) or findings (e.g. immune response).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 3 years
  The occurrence of adverse events from injection to Day 1095 (36 months/three years, in all participants, in all groups:

SECONDARY OUTCOMES:
Immunogenicity | 6 months
  Evaluate the immunogenicity of influenza antigens contained in TIV when combined with PAL adjuvant as measured by haemagglutination inhibition (HAI) titres, pre-injection (Day 0) and post-injection (Days 28, 120 and 180).
Immunogenicity of TIV combined with PAL | 6 months
  Immunogenicity of the influenza antigens contained in TIV when combined with PAL adjuvant as measured by IgG and IgG1 antibody directed to influenza A viral nucleoproteins on Days 0, 28, 120 and 180.
Immune responses | 6 months
  Describe cellular immune responses to the investigational products as assessed by antigen-secreted interferon-gamma secretion, and interferon-gamma to IL-10 ratio, pre-injection (Day 0) and post-injection (Day 28, Day 120 and Day 180).
Induced immune responses | 6 months
  Describe immune responses induced by PAL adjuvant combined with TIV as measured by Granzyme B levels in Peripheral Blood Mononuclear Cells (PBMC), pre-injection (Day 0) and post-injection (Day 28, Day 120 and Day 180).
Solicited and General Adverse Events | up to 6 months
  The occurrence of each solicited local and general AE (adverse event), during a 7-day follow-up period after injection (i.e. the day of injection and 6 subsequent days).
Hematological laboratory values | up to 6 months
  The occurrence of any hematological (hemoglobin level, WBC (white blood cells), lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (ALT, AST(angiotensin sensitivity test) and creatinine) laboratory abnormality at Day 0 and at Day 7.
Unsolicited Adverse Events | 3 years
  The occurrence of any unsolicited AE, during a 28-day follow-up period after injection (i.e. the day of injection and 27 subsequent days), and through to Day 1095. The occurrence of any SAE through to Day 1095.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Langley, M.D., Principal Investigator — Canadian Center for Vaccinology
Locations (1):
- Canadian Center for Vaccinology, Halifax, Nova Scotia, Canada